CLINICAL TRIAL: NCT05936983
Title: Comparison of Physical Fitness, Physical Activity Level, Depression and Quality of Life in Patients With Bipolar Disorder and Schizophrenia With Healthy Controls
Brief Title: Comparison of Physical Fitness, Physical Activity Level in Patients With Bipolar Disorder and Schizophrenia
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/514/247/4
Record Dates: First submitted 2023-05-31; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Bipolar disorder: Participants will be asked to fill out a structured questionnaire containing their sociodemographic characteristics. Then, Anthropometric Measurements, Eurofit test battery, Rapid Depressive Symptom Inventory-Self-Report Form and International physical activity questionnaire will be applied respectively.
- Patients with Schizophrenia group: Participants will be asked to fill out a structured questionnaire containing their sociodemographic characteristics. Then, Anthropometric Measurements, Eurofit test battery, Rapid Depressive Symptom Inventory-Self-Report Form and International physical activity questionnaire will be applied respectively.
- Healthy group: Participants will be asked to fill out a structured questionnaire containing their sociodemographic characteristics. Then, Anthropometric Measurements, Eurofit test battery, Rapid Depressive Symptom Inventory-Self-Report Form and International physical activity questionnaire will be applied respectively.

SUMMARY:
According to the World Health Organization; Bipolar disorder ranks in the top 20 causes of disability among all medical conditions and 6th among mental disorders worldwide. Bipolar disorder is noted as a serious mental illness involving emotional ups and downs.

DETAILED DESCRIPTION:
Schizophrenia is a chronic mental disorder characterized by the appearance of both positive symptoms such as hallucinations and delusions and negative symptoms such as apathy and withdrawal, repetition of cognitive skills, and disorganization. In this study, it was aimed to compare physical fitness, physical activity level, depression and quality of life in bipolar disoder and schizophrenic patients with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with bipolar disorder and schizophrenia by a physician according to DSM-5 criteria

  * Individuals with bipolar and schizophrenia between the ages of 30-55
  * Patients without any other accompanying psychiatric disorder
  * Patients who can communicate
  * Patients who agreed to participate in this study and gave informed consent

Exclusion Criteria:

* Patients with a psychiatric diagnosis other than bipolar and schizophrenia.
* Pregnancy condition
* Those who did not consent to participate in the study

Ages: 30 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: patients with Bipolar disorder and schizophrenia come to the community mental health center regularly
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Waist measurement - Antropometric Measurements | 4 weeks
  Waist measurement is measured from the narrowest area between the subcostal region and the iliac crest.
Abdomen measurement - Antropometric Measurements | 4 weeks
  Abdomen measurement is measured at the level of the umbilicus without compression of the tissues.
The hip measurement - Antropometric Measurements | 4 weeks
  The hip measurement is measured from the thickest part of the hip area.
Eurofit Test Battery | 4 weeks
  A test-retest design was applied to test the reproducibility of several Eurofit test battery items. Supervision and measurement of the Eurofit test battery was performed by one trained mental health physical therapist following a standardized procedure. The Eurofit test battery included seven items and involved the assessment of the following measures: whole body balance, speed of limb movement, flexibility, explosive strength, static strength, abdominal muscular endurance and running speed.
Quick Inventory of Depressive Symptomatology (QIDS-SR16) scale | 4 weeks
  QIDS-SR consists of 16 items each ranging from 0 to 3. It is scored by summing the highest response in each of a set of questions relating to sleep, weight and psychomotor symptoms and then adding the remaining items
International Physical Activity Questionnaire | 4 weeks
  The IPAQ questionnaires list activities and request estimates of durations and frequencies for each activity engaged in over the past week. Durations are multiplied by known METs per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores. A sitting question is not included in physical activity score.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Akbuğa Koç, Principal Investigator — Yeditepe University; İsmail Koç, Principal Investigator — Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No